CLINICAL TRIAL: NCT03323801
Title: A Pilot Trial of 13-cis Retinoic Acid (Isotretinoin) for the Treatment of Men With Azoospermia
Brief Title: RA-4: 13-cis Retinoic Acid for Treatment of Men With Azoospermia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, John Amory, Professor, School of Medicine, General Internal Medicine, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001055; K24HD082231 (NIH)
Record Dates: First submitted 2017-10-24; First posted 2017-10-27 (Actual); Results first posted 2021-10-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-09

CONDITIONS: Male Infertility, Azoospermia
Keywords: Infertility
MeSH Terms: conditions — Infertility, Male; Azoospermia; Infertility | interventions — Isotretinoin

STUDY DESIGN:
Intervention Model Description: 20 mg 13-cis retinoic acid twice daily (BID) with meals for 32 weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 13-cis retinoic acid (Experimental): 20 mg 13-cis retinoic acid twice daily (BID) with means for 32 weeks
  Interventions: Drug: 13-cis retinoic acid

INTERVENTIONS:
Drug: 13-cis retinoic acid — Accutane is used for the treatment of severe acne
  Other Names: Accutane, Isotretinoin

SUMMARY:
Men with infertility and normal hormone levels have few options for fertility treatment. Previous research suggests that men with infertility may have low levels of the active form of Vitamin A, called retinoic acid, in their testes. In a pilot study of 20 men with low numbers of sperm (<10 million motile sperm), roughly half the men showed improvement in sperm production. Thus, we want to see if retinoic acid administration to men with azoospermia (no sperm present) can initiate sperm production.

DETAILED DESCRIPTION:
Twenty men with infertility, aged 21 - 60, due to azoospermia (no apparent sperm in the ejaculate on two separate occasions) will be enrolled in a single-arm pilot trial of daily oral therapy of 20 mg twice daily of 13-cis retinoic acid for 32 weeks. The impact of treatment on the appearance of sperm in the ejaculate will be determined by monthly semen analyses.

Note: The outcome measure of serum and seminal plasma 13-cis-retinoic acid concentrations was entered in error and not intended to be reported for this study. Information on these levels is available in our earlier study of 13-cis-retinoic acid in men with sub-fertility. Amory et al. Andrology 2017 5:1115-1123.

ELIGIBILITY:
Inclusion Criteria: Infertile men with azoospermia on at least two semen analyses separated by at least one week, and no pregnancy with partner with normal cycles and normal hysterosalpingogram despite >1 year of unprotected intercourse.

-

Exclusion Criteria: hypogonadotropic hypogonadism (that might respond to gonadotropin injections); use of anabolic steroids,illicit drugs, or consumption of more than 4 alcoholic beverages daily; current therapy with retinoic acid (eg Accutane) or vitamin A- of use of isotretinoin within eight weeks of start of dosing;phenytoin, or medication containing tetracycline; personal history of serious psychiatric disorders, score of greater than 15 on the PHQ9 (mood) questionnaire; elevated serum serum triglycerides or other abnormal serum chemistry values; history of inflammatory bowel disease or bone disease; not living within catchment area; participation in another clinical trial

-

Ages: 21 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2019-05-16 (Actual); Study Completion 2019-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John K Amory, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States

REFERENCES:
- [Background] Jequier AM, Holmes SC. Primary testicular disease presenting as azoospermia or oligozoospermia in an infertility clinic. Br J Urol. 1993 Jun;71(6):731-5. doi: 10.1111/j.1464-410x.1993.tb16075.x. PMID 8102079
- [Background] de Kretser DM. Male infertility. Lancet. 1997 Mar 15;349(9054):787-90. doi: 10.1016/s0140-6736(96)08341-9. No abstract available. PMID 9074589
- [Background] Schlegel PN. Nonobstructive azoospermia: a revolutionary surgical approach and results. Semin Reprod Med. 2009 Mar;27(2):165-70. doi: 10.1055/s-0029-1202305. Epub 2009 Feb 26. PMID 19247918
- [Background] Napoli JL. Retinoic acid: its biosynthesis and metabolism. Prog Nucleic Acid Res Mol Biol. 1999;63:139-88. doi: 10.1016/s0079-6603(08)60722-9. PMID 10506831
- [Background] Doyle TJ, Braun KW, McLean DJ, Wright RW, Griswold MD, Kim KH. Potential functions of retinoic acid receptor A in Sertoli cells and germ cells during spermatogenesis. Ann N Y Acad Sci. 2007 Dec;1120:114-30. doi: 10.1196/annals.1411.008. Epub 2007 Sep 28. PMID 17905941
- [Background] Koubova J, Menke DB, Zhou Q, Capel B, Griswold MD, Page DC. Retinoic acid regulates sex-specific timing of meiotic initiation in mice. Proc Natl Acad Sci U S A. 2006 Feb 21;103(8):2474-9. doi: 10.1073/pnas.0510813103. Epub 2006 Feb 6. PMID 16461896
- [Background] Anderson EL, Baltus AE, Roepers-Gajadien HL, Hassold TJ, de Rooij DG, van Pelt AM, Page DC. Stra8 and its inducer, retinoic acid, regulate meiotic initiation in both spermatogenesis and oogenesis in mice. Proc Natl Acad Sci U S A. 2008 Sep 30;105(39):14976-80. doi: 10.1073/pnas.0807297105. Epub 2008 Sep 17. PMID 18799751
- [Background] Chung SS, Wang X, Wolgemuth DJ. Expression of retinoic acid receptor alpha in the germline is essential for proper cellular association and spermiogenesis during spermatogenesis. Development. 2009 Jun;136(12):2091-100. doi: 10.1242/dev.020040. PMID 19465599
- [Background] Dufour JM, Kim KH. Cellular and subcellular localization of six retinoid receptors in rat testis during postnatal development: identification of potential heterodimeric receptors. Biol Reprod. 1999 Nov;61(5):1300-8. doi: 10.1095/biolreprod61.5.1300. PMID 10529278
- [Background] Lohnes D, Kastner P, Dierich A, Mark M, LeMeur M, Chambon P. Function of retinoic acid receptor gamma in the mouse. Cell. 1993 May 21;73(4):643-58. doi: 10.1016/0092-8674(93)90246-m. PMID 8388780
- [Background] Lufkin T, Lohnes D, Mark M, Dierich A, Gorry P, Gaub MP, LeMeur M, Chambon P. High postnatal lethality and testis degeneration in retinoic acid receptor alpha mutant mice. Proc Natl Acad Sci U S A. 1993 Aug 1;90(15):7225-9. doi: 10.1073/pnas.90.15.7225. PMID 8394014
- [Background] Ghyselinck NB, Vernet N, Dennefeld C, Giese N, Nau H, Chambon P, Viville S, Mark M. Retinoids and spermatogenesis: lessons from mutant mice lacking the plasma retinol binding protein. Dev Dyn. 2006 Jun;235(6):1608-22. doi: 10.1002/dvdy.20795. PMID 16586441
- [Background] Hoting VE, Schutte B, Schirren C. [Isotretinoin treatment of acne conglobata. Andrologic follow-up]. Fortschr Med. 1992 Aug 20;110(23):427-30. German. PMID 1398387
- [Background] Vogt HJ, Ewers R. [13-cis-Retinoic acid and spermatogenesis. Spermatological and impulse cytophotometric studies]. Hautarzt. 1985 May;36(5):281-6. German. PMID 3159708
- [Background] Torok L, Kadar L, Kasa M. Spermatological investigations in patients treated with etretinate and isotretinoin. Andrologia. 1987 Nov-Dec;19(6):629-33. doi: 10.1111/j.1439-0272.1987.tb01915.x. PMID 3481225
- [Background] Nya-Ngatchou JJ, Arnold SL, Walsh TJ, Muller CH, Page ST, Isoherranen N, Amory JK. Intratesticular 13-cis retinoic acid is lower in men with abnormal semen analyses: a pilot study. Andrology. 2013 Mar;1(2):325-31. doi: 10.1111/j.2047-2927.2012.00033.x. Epub 2012 Nov 29. PMID 23413144

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 13-cis Retinoic Acid
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Men with infertility due to azoospermia
Arm/Group | 13-cis Retinoic Acid
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 36 [31 to 42]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Total Motile Sperm
Description: Number of participants with undetectable or detectable sperm in their ejaculates.
Time Frame: up to 32 weeks
Population: Men had idiopathic azoospermia, without evidence of obstruction or know genetic causes of azoospermia, although one man had known AZFc deletion
Measure: Count of Participants; unit: Participants
Groups:
- Accutane-13-cis Retinoic Acid: 20 mg 13-cis retinoic acid twice daily (BID) with means for 32 weeks
  13-cis retinoic acid: Accutane is used for the treatment of severe acne
Arm/Group | Accutane-13-cis Retinoic Acid
Number analyzed (Participants) | 9
Participants
  undetectable | 8
  detectable motile sperm | 1

2. Primary Outcome: Total Sperm and Percentage of These Sperm That Were Motile
Description: Number of total sperm in ejaculate and percentage of these sperm that were motile
Time Frame: 32 weeks
Population: Only man who developed sperm in ejaculate on treatment
Measure: Number; unit: Percent of sperm that were motile
Units Other Than Participants: Total sperm in the ejaculate
Arm/Group | 13-cis Retinoic Acid
Number analyzed (Participants) | 1
Number analyzed (Total sperm in the ejaculate) | 32500
Percent of sperm that were motile | 20

3. Secondary Outcome: Serious and Non-Serious Adverse Effects
Description: Number of participants with Serious and Non-Serious Adverse effects associated with treatment with 13-cis retinoic acid
Time Frame: 32 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Accutane-13-cis Retinoic Acid
Number analyzed (Participants) | 10
Participants | 1

ADVERSE EVENTS:
Time Frame: 32 weeks
Arm/Group | Accutane-13-cis Retinoic Acid
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 1/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Accutane-13-cis Retinoic Acid (N=10)
nephrotic syndrome (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Accutane-13-cis Retinoic Acid (N=10)
cramps (Musculoskeletal and connective tissue disorders) | 1 (1) — Muscle cramps

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-01-12): https://cdn.clinicaltrials.gov/large-docs/01/NCT03323801/Prot_SAP_002.pdf
  • Informed Consent Form (2017-05-23): https://cdn.clinicaltrials.gov/large-docs/01/NCT03323801/ICF_001.pdf